CLINICAL TRIAL: NCT07105436
Title: Utility of the Thopaz+ System in Evaluating Persistent Air Leaks
Brief Title: Thopaz for PALs Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Kai Swenson (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Kai Swenson, Instructor in Medicine, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Other Study IDs: 2024P001113
Record Dates: First submitted 2025-06-18; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Persistent Air Leaks
Keywords: Persistent Air Leaks; Chest Tube; Waterseal; Thopaz+

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Persistent air leak quantification — In this trial, patients with PALs will have their chest tubes connected to the Thopaz+ system. The Thopaz+ will continuously quantify the volume of air leaks, providing real-time data for analysis.
  Data from both the Thopaz+ and standard serial occlusion test with Fogarty balloon will be combined and integrated to provide a comprehensive assessment of the air leak source. The bronchoscopic will perform standard visual assessment of changes in air leak during serial balloon occlusion in order to identify the best region for endobronchial treatments; use of measurements from the Thopaz and serial balloon occlusion test will be allowed as part of clinical reasoning but are not required to be used by the treating clinician.

SUMMARY:
Persistent air leaks (PALs) are a common postoperative complication resulting from tears in the visceral pleura or peripheral lung resections. Although highly prevalent with significant consequences, traditional assessment methods lack the capability to objectively quantify air leaks, which further complicates management, results in inconsistent decision making, and prolongs hospital stays. By incorporating the Thopaz+ system, the investigators can introduce a reliable approach to objectively quantify air leaks, potentially improving clinical outcomes.

The purpose of this protocol is to perform a pilot prospective controlled clinical trial to evaluate the utility of incorporating the Thopaz+ system and its volume quantification ability in evaluating patients with persistent air leaks (PALs) to guide treatment decisions, specifically endobronchial valves (EBVs).

In the targeted cohort, the Thopaz+ will be connected to the chest tube and the data collected will be combined with that of serial balloon occlusion testing with a Fogarty balloon to accurately localize the air leak source, and subsequently consider the correct placement of EBVs. The investigators will thereby determine whether this experimental strategy will yield a more accurate and objective assessment of air leaks, facilitating timely interventions and improved patient outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a prospective controlled clinical trial. The investigators' target demographic includes all adult patients with lung resection and/or non-lung resection-related PAL with ipsilateral chest tubes who were not candidates for surgical intervention or patients who refused the intervention. These patients would undergo a multidisciplinary review by thoracic surgery, interventional pulmonary and the primary care team to consider a bronchoscopic approach with endobronchial valves and possibly bronchial blood patch, which is currently considered standard of care at our institution. During this standard-of-care intervention, quantitative assessment of distal occluded airway pressures/flows in various airways, as well as quantitative assessment of air leak volume will be assessed.

In current medical practice, when EBVs are considered in the context of managing PALs, bronchoscopists may opt to either conduct complete lobar occlusion (sealing of all segments within the target lobe) or segmental occlusion (sealing only selected segments within the target lobe). The decision is usually guided by localizing the source of air leak which is usually done by monitoring the reduction of air leak on the pleural drainage device following serial inflation of a Fogarty Catheter at various locations within the endobronchial tree and monitoring change in air leak visually in the pleural drainage system.

In this trial, patients with PALs will have their chest tubes connected to the Thopaz+ system. The Thopaz+ will continuously quantify the volume of air leaks, providing real-time data for analysis.

Data from both the Thopaz+ and standard serial occlusion test with Fogarty balloon will be combined and integrated to provide a comprehensive assessment of the air leak source. The bronchoscopist will perform standard visual assessment of changes in air leak during serial balloon occlusion in order to identify the best region for endobronchial treatments; use of measurements from the Thopaz and serial balloon occlusion test will be allowed as part of clinical reasoning but are not required to be used by the treating clinician.

Continuous monitoring using the Thopaz+ system may continue post-procedure to track changes in air leak volumes and patient recovery, ensuring timely interventions and optimal patient outcomes. This integrated approach aims to provide a more accurate, objective, and efficient method of managing PALs compared to traditional techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalized with a persistent air leak (PAL) lasting ≥5 days despite continuous chest tube drainage.
* Undergoing bronchoscopy as part of clinical care for PAL management.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Contraindications to bronchoscopy or EBV placement.
* Pregnancy.
* Inability to tolerate general anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects will be patients who meet the inclusion criteria including a willingness to read, understand, and sign the informed consent. Recruitment of study subjects will be from the pool of admitted patients from our inpatient service. They will be recruited in a consecutive fashion from the clinical practices of the investigators from BIDMC.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Successful Intraoperative Quantification of Air Leak Volume Using Thopaz+ Digital Drainage System | During procedure
  Feasibility will be defined by the ability to obtain continuous, interpretable quantitative air leak volume data (in mL/min) during bronchoscopic evaluation of persistent air leaks. Successful quantification is defined as capturing measurable air leak volume data during serial balloon occlusion in at least one airway segment. The outcome will be reported as the number and percentage of participants with successful measurements out of the total enrolled population.

SECONDARY OUTCOMES:
Percentage of patients with identifiable lobar or segmental airways responsible for PAL | During procedure
  Percentage of patients with identifiable lobar or segmental airways responsible for PAL
Maximum decrease in volume of air leak during serial balloon occlusion, as measured by Thopaz+ device | During procedure
Treatment success: decrease of one grade in Cerfolio classification for air leaks or removal of continuous suction from chest drain. | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
  The Cerfolio classification categorizes air leaks based on their occurrence during the respiratory cycle, with grades 1-4 indicating increasing severity. Grade 1 is a forced expiratory leak, seen during coughing; Grade 2, expiratory; Grade 3, inspiratory; and Grade 4, continuous during both inspiration and expiration
Treatment failure: no decrease in the degree of the air leak (Cerfolio classification) and the need for continuous suction for chest drain | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
Length of stay following EBV placement | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
Duration of chest tube following bronchoscopy | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
Change in Air Leak Severity Graded by Cerfolio Classification | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
  The Cerfolio classification categorizes air leaks based on their occurrence during the respiratory cycle, with grades 1-4 indicating increasing severity. Grade 1 is a forced expiratory leak, seen during coughing; Grade 2, expiratory; Grade 3, inspiratory; and Grade 4, continuous during both inspiration and expiration
Change in Quantitative Air Leak Volume Measured by Thopaz+ Digital Drainage System | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
  The Thopaz+ device will be used to continuously measure the volume of air leak (in mL/min) before and after bronchoscopic intervention. The outcome will report the change in air leak volume from baseline (pre-bronchoscopy) to post-bronchoscopy values.
The need for additional non-surgical intervention | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)
The need for additional surgical intervention for PAL such as video-assisted thoracoscopic surgery with mechanical pleurodesis, blebectomy or lobectomy | From enrollment until 8 weeks follow-up (as per standard of care for bronchoscopic treatment of PALs)